CLINICAL TRIAL: NCT06461403
Title: Inhaler Trainer Efficacy Study: Interactive Training Tool Providing Technique Feedback for COPD/Asthma Medication Delivery
Brief Title: Inhaler Trainer Efficacy Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Koronis Biomedical Technologies (Industry)
Collaborators: University of Chicago (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB21-1418; 5R44AG071430 (NIH)
Record Dates: First submitted 2024-04-12; First posted 2024-06-17 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-08

CONDITIONS: Asthma; Copd; Acute Exacerbation of COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Inhaler Trainer Device (Experimental): The Inhaler Trainer Device will monitor patients' inspiratory waveform to confirm technique compliance based on objective metrics and provide feedback on how to better perform technique. This intervention utilizes an instrumented training inhaler capable of accurately measuring the real-time inspiratory airflow achieved by the user when they perform their inhale maneuver. If a user's inspiratory flow fails to produce an inspiratory waveform with sufficient airflow parameters, the inhaler device may not optimally aerosolize the medication, and the delivered dosage to the lung will be negatively affected. The device measures the most important flow parameters in the users' real-time inspiration performance and translates them into an estimation of the dose delivered to the lung, based on detailed characterization of the user's inhaler product.
  Interventions: Device: Inhaler Trainer System; Other: Initial Inhaler Use Assessment; Other: Inhaler Use Instruction
- Brief Interventions (BI) (Active Comparator): During inpatient admission, participants randomized to the BI condition will receive the following: First, they will undergo an initial assessment of their respiratory inhaler technique using device-specific checklists. Participants will then be given step-by-step verbal instructions and a copy of written instructions by the trained educator describing appropriate inhaler technique for their respiratory inhalers. The educator will not demonstrate the appropriate use of each inhaler to the patient, though the educator will be free to answer questions about appropriate use if posed by the study subject.
  Interventions: Other: Initial Inhaler Use Assessment; Other: Inhaler Use Instruction

INTERVENTIONS:
Device: Inhaler Trainer System — The system consists of an instrumented training inhaler capable of accurately measuring the real-time inspiratory airflow achieved by the user when they perform their inhale maneuver. The inhaler trainer system consists of a detachable/disposable mouthpiece and a reusable electronics module. The electronics module measures flow/pressure achieved by the patient and wirelessly transmits this data to a PC. The PC software analyzes the real-time inhalation flow data to enable the monitoring of the following quantities: Flow Rate, Duration, and Maximum Pressure Slope. These quantities will be used in the computation of the assessment metric, providing the user with real-time feedback about their inhalation technique. In addition, the software includes features to support the human study and provides fully functional inhaler education features for the expert test evaluators.
  Arms: Inhaler Trainer Device
Other: Initial Inhaler Use Assessment — Patients will undergo an initial assessment of their respiratory inhaler technique for their respiratory inhaler devices using device-specific checklists
Other: Inhaler Use Instruction — Participants will then be given step-by-step verbal instructions and a copy of written instructions by the trained educator describing appropriate inhaler technique for their respiratory inhalers.

SUMMARY:
This will be a randomized, controlled, clinical trial. The investigators aim to determine the feasibility of and efficacy of the Inhaler Trainer Device for ongoing inhaler skill training.

The research team will enroll 140 patients from the inpatient or outpatient setting from the University of Chicago Medicine over the course of up to 12 months. Participants will complete assessments, a lung function test via spirometry, and inhaler education via either the Inhaler Trainer Device learning program or Brief Intervention.

All participants will return at 6 weeks (window of +/- one week) post-initial inhaler education for an in-person evaluation of their inhaler skills, lung function, and acute care utilization. Finally, a post-study semi-structured interview will be conducted to gather feedback on the device after the 6-week visit has been completed.

DETAILED DESCRIPTION:
The research team will enroll 140 patients from the inpatient or outpatient setting from the University of Chicago Medicine inpatient services, COPD/APN clinic, general medicine clinic, and/or Pulmonary clinic until all participants have been enrolled (approximately over the course of 12 months).

Patients will be randomized into one of two treatment conditions: one including use of the inhaler training device and one with our standard brief intervention.

After obtaining informed consent, participants will complete assessments, including a lung function test via spirometry, and inhaler education via either the Inhaler Trainer Device learning program or standard education techniques. Participants randomized to the inhaler training device arm will be trained on how to use their inhaler and the inhaler trainer device. The Inhaler Trainer Device will monitor the patient's inspiratory waveform to confirm technique compliance based on objective metrics and provide feedback on how to better perform technique.

Participants will continue to use their inhaled medications with the inhaler trainer device for 6 weeks post-baseline. They will return at 6 weeks post-initial instruction for an in-person evaluation of their inhaler skills, lung function, and acute care utilization. Finally, a post-study semi-structured interview will be conducted to gather feedback on the device after the 6-week visit has been completed. This interview will occur either during the 6-week follow-up visit or at a later time via phone call or zoom call. In the interview, a standard elicitation framework guided by the Integrative Model (IM) of Behavioral Prediction and Change will be used to generate feedback on training experience. The research team will also prompt participants to give feedback on the design, content, and functionality of the inhaler and training system. Additional prompts and questions will be used to ensure that information is provided that speaks to participants' perceptions of the positive and negative consequences related to using the trainer.

The statistical team at the University of Chicago will conduct analyses including descriptive summaries using means, medians, proportions, scatterplots, and histograms to describe the data. McNemar's chi-squared tests will be used to compare 30-day follow-up and inhaler misuse (≤10/12 steps correct) post-education vs. baseline. To model over time, we will use generalized linear mixed method (GLMM) or generalized estimating equations (GEE). A two-tailed p-value less than 0.05 will define statistical significance. The sample size was powered on the primary outcome in Aim 1 for difference in correct MDI use (>75% steps correct) between baseline and at 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85
* Physician diagnosis of COPD or asthma
* Has been prescribed or is being prescribed one of the inhalers listed below (DPI inhaler product, Active pharmaceutical ingredient):

  1. Serevent®Diskus®(GSK), Salmeterol
  2. Incruse Ellipta (GSK), Umeclidinium
  3. Spiriva Handihaler (BIP),Tiotropium
  4. Tudorza Pressair (AstraZeneca), Aclidinium
* Inexperienced with inhaler trainer device (defined by never having had inhaler training using an auxiliary tool besides an actual inhaler and spacer)

Exclusion Criteria:

* Physician declines to provide assent
* Patient unable to provide consent (e.g., history of cognitive impairment, unable to understand English) or declines to provide consent
* Does not meet inclusion criteria

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Inhaler technique assessment | 6 weeks
  Participants' overall inhaler technique will be scored via observation by a trained research educator. This assessment will follow a validated checklist and scoring system based the inhaler the patient is using. For example, if the patient is using a Spiriva handihaler, each of the following steps will be marked as either complete or incomplete: removes cap of inhaler and spacer, shakes inhaler up and down, attaches inhaler to spacer, breathes out fully, breathes out away from spacer/MDI, closes lips around spacer mouthpiece, presses down on canister one time, breathes in slowly, holds breath for at least five seconds, removes spacer from mouth before breathing normally, breathes normally for at least 30-60 seconds, repeats steps 2-11 for second puff. There will be a designated spot for any qualitative findings identified by the educator. Scores will be compared to baseline and post-training results at 6 weeks post-inhaler technique training.

SECONDARY OUTCOMES:
Estimated inhaled dosage | 6 weeks
  Estimated inhaled dosage is estimated by the prototype training device and is used to inform the training session. Dosage will be compared to the baseline and training session. Dosage will be compared to the baseline and training session results at 6 weeks post inhaler technique training.
Usability | 6 weeks
  To assess the overall usability and acceptability of the system, a short Likert-type usability survey will be developed based on the system usability scale and tailored to their inhaler type. For example, participants may be asked on a scale from 1-5, to what degree they agree to statements similar to "I thought the training system was easy to use", with 1 being strongly disagree, and 5 being strongly agree. Participants will complete the assessment, which will be administered by a trained interviewer.
Spirometer pulmonary function measures | 6 weeks
  Forced Expiratory Volume in One Minute (FEV1). Scores will be compared to baseline at 6 weeks post inhaler technique training.
Spirometer pulmonary function measure: FVC | 6 weeks
  Forced Vital Capacity (FVC). Scores will be compared to baseline at 6 weeks post inhaler technique training.
Spirometer pulmonary function measure: PEF | 6 weeks
  Peak Expiratory Flow (PEF). Scores will be compared to baseline at 6 weeks post inhaler technique training.
Inhalation Parameters - flow slope | 6 weeks
  Flow slope will be measured by the prototype trainer device and compared to the baseline and training session at 6 weeks post inhaler technique training.
Inhalation Parameters - peak flow | 6 weeks
  Peak flow will be measured by the prototype trainer device and compared to the baseline and training session at 6 weeks post inhaler technique training.
Inhalation Parameters - total volume | 6 weeks
  Total volume will be measured by the prototype trainer device and compared to the baseline and training session results at 6 weeks post inhaler technique training.
Symptom Control: mMRC | 6 weeks
  Symptoms will be assessed with the mMRC(Modified Medical Research Counsel dyspnea scale assessment), a validated tool that stratifies severity of dyspnea in respiratory diseases, particularly COPD. It is often used to establish baseline functional impairment due to dyspnea attributable to respiratory disease. The minimum value from this tool is 0, which indicates that the patient "only gets breathless with strenuous exercise". The maximum value of the tool is 4, which indicates that the patient "is too breathless to leave the house or is breathless when dressing". Results will be compared to the baseline and training session results at 6 weeks post inhaler technique training.
Symptom Control: Modified Borg Dyspnea Scale | 6 weeks
  Symptoms will be assessed with the Modified Borg Dyspnea Scale. The minimum value of this tool is 0, which indicates that the patient experiences no shortness of breath. The maximum value of this tool is 10, which indicates that the patient is experiencing very severe shortness of breath. Results will be compared to the baseline and training session results at 6 weeks post inhaler technique training.
Symptom control: Asthma | 6 weeks
  Asthma symptoms will be measured by the following assessments: ASSI (Asthma Symptom Severity Index). Patients will give a number in response to the question: "How is your asthma/COPD right now?" from 0 - 10, with 0 indicating no symptoms, and 10 indicating maximal symptoms. Results will be compared to the baseline and training session results at 6 weeks post inhaler technique training.
Disease control: COPD | 6 weeks
  COPD disease control will be measured with the CAT (COPD Assessment Test), which is a questionnaire for people with COPD that is designed to measure the impact of COPD on a person's life. The questionnaire is composed of 8 statements/questions with which the patient responds on a 0-5 scale. Total scores for the questionnaire can range from 0 - 40, with 0 indicating well controlled COPD and 40 indicating extremely poorly controlled COPD. Results will be compared to the baseline and training session results at 6 weeks post inhaler technique training.
Disease control: Asthma | 6 weeks
  Asthma control will be measured with the asthma control questionnaire. This questionnaire measures the adequacy of asthma control and change in asthma control that occurs either spontaneously or as a result of treatment. It is a 20 item questionnaire surveying effects of breathing problems on patients' everyday life. There are two sections to the questionnaire. The first 13 questions have answers ranging from 1-3, (1 = YES, 2 = NO, and 3 = N/A). The last 7 questions have answers ranging from 1-4 (1 = YES, 2 = NO, 3 = UNABLE, 4 = N/A). Results will be compared to the baseline and training session results at 6 weeks post inhaler technique training.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Koronis Biomedical Technology researchers and our collaborative research partners at the University of Chicago are active contributors to a variety of peer-reviewed publications, academic conference venues, and industrial consortiums. A wide variety of research conclusions stemming from the proposed project will be submitted for public disclosure through these various venues. We aim to spur improvements to COPD/asthma and COPD/asthma disease management options worldwide.
  It is our express intention to participate in the research endeavor of the larger research community and we have several strategies to explicitly share our data, insight and analysis tools while maintaining subject confidentiality. We intend to broadly disseminate our insights through prompt and complete publication in peer-reviewed journals.
  Additionally, Koronis Biomedical Technologies will adopt the NIH Policy for dissemination of NIH-Funded Clinical trial information, published in full as NOT-OD-16-149.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code